CLINICAL TRIAL: NCT05854277
Title: Inception, Validation and Clinical Utility of a Score to Assess the Completeness of Caecal Visualisation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: BC-09013
Record Dates: First submitted 2023-03-15; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Colonic Polyp; Colorectal Cancer
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopists (Other)
  Interventions: Other: educational video

INTERVENTIONS:
Other: educational video — To explain the novel score, a six-minute instructional video was compiled and available to watch, as well as an online tool on the GIEQs website that could be used to grade the image-sets using the score.

SUMMARY:
CCIS is a novel score, created specifically to evaluate the completeness of caecal visualized. It can be applied to a single or multiple images. To create the CCIS, the caecum was divided into eight parts: the appendiceal orifice (AO), the tri-radiate fold part 1 (TF-1), 2 (TF-2), 3 (TF-3) and four outer quadrants (OQ 1-4). The ileo-caecal valve (ICV) is a reference point but is not part of the score. The quadrant adjacent to the ICV is labelled OQ1. The three other quadrants are labelled clockwise from this quadrant. The tri-radiate folds are also labelled clockwise with TF1 representing the triangle side that is majority-contained within OQ1. TF2 and TF3 are then labelled clockwise from TF1.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists >18 years old

Exclusion Criteria:

* Endoscopist not signing informed consent
* Any other medical doctor not connected with endoscopic practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
VALIDATE A NOVEL SCORE FOR THE COMPLETENESS OF CAECAL INTUBATION | 4 weeks
  To create the CCIS, the caecum is divided into eight parts: the appendiceal orifice (AO), the tri-radiate fold part 1 (TF-1), 2 (TF-2), 3 (TF-3) and four outer quadrants (OQ 1-4). The ileo-cacecal valve (ICV) is a reference point but is not part of the score. The quadrant adjacent to the valve is labelled OQ1. The three other quadrants are labelled clockwise from this quadrant. For every component of the CCIS that is completely visualized on the image, one point is gained with a maximum possible CCIS of 8 and a minimum of 0. Participants were asked to answer the same six questions for each image-set.
  * Is this an image of the caecum?
  * What is the Boston Bowel Preparation score for this segment of the colon?
  * What is your subjective first impression (yes/no) regarding completeness of caecal intubation?
  * What subjective percentage do you believe was assessed?
  * What is the CCIS score for this image-set?
  * Using the online tool, which components of the CCIS were seen

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Gent, Ghent, Belgium